CLINICAL TRIAL: NCT01765023
Title: An Open-label, Fixed-sequence Study to Evaluate Pharmacokinetic Interactions Between Atorvastatin and Metformin in Healthy Male Subjects
Brief Title: Pharmacokinetic Interactions Between Atorvastatin and Metformin in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: HK inno.N Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CJ_ATM_101
Record Dates: First submitted 2012-12-12; First posted 2013-01-10 (Estimated); Last update posted 2013-04-09 (Estimated); Status verified 2013-04

CONDITIONS: Healthy
MeSH Terms: interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part A (Experimental): single administration : atorvastatin 40mg, qd, 7days(oral) combination administration : atorvastatin 40mg and metformin XR 1000mg, qd, 7days(oral)
  Interventions: Drug: Period I : atorvastatin, Period II : atorvastatin and metformin
- Part B (Experimental): single administration : metformin XR 1000mg, qd, 7days(oral) combination administration : atorvastatin 40mg and metformin XR 1000mg, qd, 7days(oral)
  Interventions: Drug: Period I : metformin, Period II : atorvastatin and metformin

INTERVENTIONS:
Drug: Period I : atorvastatin, Period II : atorvastatin and metformin
  Arms: Part A
Drug: Period I : metformin, Period II : atorvastatin and metformin
  Arms: Part B

SUMMARY:
The purpose of the study is to assess the pharmacokinetic interactions between atorvastatin and metformin single or co-administered in healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

1. Willing to adhere to protocol requirements and sign a informed consent form
2. Healthy male volunteers who are in age range of 20-55 years and the weight range is not exceed ±20% of ideal weight. Ideal weight = [height -100]*0.9
3. Subjects with no history of any significant chronic disease
4. Judged to be in good health on the basis of their vital sign, ECG, physical exam and routine laboratory data for this trial by investigators

Exclusion Criteria:

1. Subjects taking inducer or inhibitor of drug metabolism enzyme such as barbital within 28days prior to study medication dosing
2. Subjects with Symptoms of acute disease within 28days prior to study medication dosing
3. Subjects with a history of gastrointestinal diseases which might significantly change ADME of medicines
4. Subjects with a history of abdominal surgery within food and water limit
5. Subjects with a history of clinically significant allergies including drug allergies
6. Subjects with anaphylaxis to atorvastatin and/or metformin
7. Subjects with a history or plan iodine radiotherapy within 28 days prior to drug administration
8. Subjects with a history of myopathy
9. Subjects with a hereditary problems, for example, galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption
10. Clinical laboratory test values are outside the accepted normal range

    * AST or ALT >1.25 times to normal range
    * Total bilirubin >1.5 times to normal range
    * Creatinine clearance <90 mL/min
11. Subjects with a history of drug, caffeine and alcohol abuse(caffeine > 5cups/day, cigarette > 10/day, alcohol > 30g/day) or have ever drank within 7 days prior to drug administration
12. Special diet known to interfere with the absorption, distribution, metabolism or excretion of drugs (especially, consumption of grapefruit juice) within 7 days prior to drug administration
13. Donated blood within 60 days prior to dosing
14. Participated in a previous clinical trial within 60 days prior to dosing
15. Subjects who have received any drugs that might confound the results of the trial based on medical judgement by investigators within 10days prior to drug administration
16. Subjects considered as unsuitable based on medical judgement by investigators

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2012-10; Primary Completion 2012-12 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
To Evaluate PK interaction of atorvastatin and metformin | Throughout the study

SECONDARY OUTCOMES:
To Evaluate PK interaction of 2-OH-atorvastatin and metformin | Throughout the study

CONTACTS AND LOCATIONS:
Locations (1):
- Inje University Pusan Paik Hospital, Busan, South Korea